CLINICAL TRIAL: NCT00967460
Title: Effect of a Physical-activity-promoting Environment on Motor Skills, Physical Activity, Quality of Life and BMI of Children in Childcare Settings (Youp'là Bouge)
Brief Title: Effect of a Physical-activity-promoting Environment on Motor Skills, Physical Activity and Quality of Life of Children in Childcare Settings
Acronym: Youp'là bouge
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Lausanne Hospitals (Other)
Collaborators: University of Lausanne (Other); University of Basel (Other); University of Zurich (Other)
Responsible Party: Jardena J Puder, MD, University of Lausanne
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 88/09
Record Dates: First submitted 2009-08-26; First posted 2009-08-27 (Estimated); Last update posted 2011-01-28 (Estimated); Status verified 2009-08

CONDITIONS: Obesity; Inactivity
Keywords: Childhood obesity; Children; Inactivity; Physical activity; Motor skills; Motor fitness; Quality of life; Nutrition; Family
MeSH Terms: conditions — Obesity; Sedentary Behavior; Pediatric Obesity; Motor Activity

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Control group: No intervention (No Intervention): No intervention, regular childcare program
- Intervention group (Experimental): Promoting unstructured spontaneous PA through an adaptation of the built environment and the provision of a supportive social environment
  Interventions: Behavioral: Lifestyle intervention

INTERVENTIONS:
Behavioral: Lifestyle intervention — Promoting unstructured spontaneous physical in childcare through an adaptation of the built environment and the provision of a supportive social environment
  Arms: Intervention group

SUMMARY:
The purpose of the study is to evaluate the effect of a project promoting unstructured spontaneous physical activity (PA) through an adaptation of the built environment and the provision of a supportive social environment of childcare centers on motor skills, physical activity, desire to move around, body mass index (BMI), quality of life and PA and behavior of the family.

DETAILED DESCRIPTION:
The study will last one school year and includes 58 childcare centers in 3 provinces (JU, NE, VD) of the French part of Switzerland.

ELIGIBILITY:
Inclusion Criteria:

* Children in selected childcare centers

Ages: 2 Years to 5 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 1764 (Actual)
Dates: Start 2009-01; Primary Completion 2010-09 (Actual); Study Completion 2010-09 (Actual)

PRIMARY OUTCOMES:
Motor skills | 1 school year

SECONDARY OUTCOMES:
Physical activity | 1 school year
Enjoyment of physical activity | 1 school year
BMI | 1 school year
Quality of life | 1 school year
Physical activity and behavior of the family | 1 school year

CONTACTS AND LOCATIONS:
Locations (3):
- Switzerland (3):
  - Ligues de la santé, Lausanne
  - University of Lausanne Hospitals, Lausanne
  - University of Lausanne, Lausanne

REFERENCES:
- [Derived] Bonvin A, Barral J, Kakebeeke TH, Kriemler S, Longchamp A, Schindler C, Marques-Vidal P, Puder JJ. Effect of a governmentally-led physical activity program on motor skills in young children attending child care centers: a cluster randomized controlled trial. Int J Behav Nutr Phys Act. 2013 Jul 8;10:90. doi: 10.1186/1479-5868-10-90. PMID 23835207